CLINICAL TRIAL: NCT06158321
Title: The Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) in Managing Individuals With Chronic Low Back Pain and Comorbid Insomnia: A Pilot Randomized Controlled Trial
Brief Title: rTMS in Managing Individuals With Chronic Low Back Pain and Comorbid Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HongKongPU_Jeremy
Record Dates: First submitted 2023-08-24; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pain; Insomnia
Keywords: Chronic low back pain; Insomnia; rTMS; RCT
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Three-arm pilot randomized controlled trial (RCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group assignment will be concealed through opaque and sealed envelopes, which will be administered by a research assistant who is not involved in the study. The envelopes will be opened after the participant consented to participate in the trial. Assessors, participants, and therapists will be blind to the allocation of rTMS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M1 or DLPFC sham stimulation (Sham Comparator): Participants will receive M1 or DLPFC sham stimulations.
  Interventions: Device: M1 or DLPFC sham stimulation
- M1 rTMS (Experimental): Participants will receive high-frequency rTMS over M1.
  Interventions: Device: M1 rTMS
- DLPFC rTMS (Experimental): Participants will receive low-frequency rTMS over DLPFC.
  Interventions: Device: DLPFC rTMS

INTERVENTIONS:
Device: M1 or DLPFC sham stimulation — Participants receiving M1 or DLPFC sham stimulations will complete the same procedures as those in the active groups. The sham coil, with the same stimulation parameters, will provide auditory and sensory effects similar to the active coil without delivering active stimulation.
  Arms: M1 or DLPFC sham stimulation
Device: M1 rTMS — The stimulation parameter of the active M1-rTMS is a 10 Hz stimulation frequency with a total of 1500 stimulation pulses.
  Other Names: Participants will receive high-frequency rTMS over M1.
  Arms: M1 rTMS
Device: DLPFC rTMS — The stimulation parameter of the active DLPFC-rTMS is a 1 Hz stimulation frequency with a total of 1500 stimulation pulses.
  Arms: DLPFC rTMS

SUMMARY:
This pilot randomized controlled trial (RCT) aims to investigate the feasibility and efficiency of delivering different rTMS protocols in individuals with CLBP and insomnia. Participants will be randomly assigned to either the primary motor cortex (M1) rTMS, the dorsolateral prefrontal cortex (DLPFC) rTMS, or sham stimulation.

DETAILED DESCRIPTION:
Sleep disturbance exacerbates pain perception, disability, and poor prognosis in individuals with chronic low back pain (CLBP). A recent systematic review demonstrated that improvements in sleep disturbance were associated with corresponding improvements in pain intensity, recovery, and disability in individuals with CLBP. These findings indicate that achieving restorative sleep is likely to mitigate chronic pain symptoms. The application of rTMS at a specific frequency over a focal brain area has been proposed as a promising treatment for chronic pain and insomnia independently. To date, no studies have compared the effectiveness of different rTMS protocols in treating comorbid CLBP and insomnia. Given the above, the current study aims to investigate the feasibility and acceptability of delivering different rTMS protocols in individuals with CLBP and insomnia and explore the relative therapeutic efficacy of these protocols on pain and sleep parameters at immediate post-treatment and one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. participants aged between18 and 65 years;
2. willing to participate in the study and randomization;
3. having stable pharmacological or nonpharmacological treatments for pain or sleep at least one month prior to study participation;
4. having CLBP (defined as pain between 12 ribs and gluteal crease with or without leg pain that has persisted for at least three months)
5. diagnosing insomnia using the Brief Insomnia Questionnaire (BIQ) based on the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5)

Exclusion Criteria

1. specific causes of CLBP (e.g., spondylosis, spondyloarthropathy, or vertebral fracture);
2. pregnancy or nursing;
3. previous spinal surgery;
4. inflammatory or autoimmune diseases;
5. other sleep disorders (e.g., sleep apnea or restless leg);
6. presence of severe psychopathologies, neurological, or physical disease directly related to the onset of insomnia (e.g., depression, substance abuse, or alcohol abuse);
7. severe dependence on hypnotic drugs;
8. concurrent receipt of new treatments outside the scope of the study;
9. contraindications to use rTMS (e.g., severe head trauma, intracranial hypertension, implanted ferromagnetic devices, history of epilepsy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate | Two weeks
  The percentage of eligible participants
Recruitment rate | Two weeks
  The percentage of eligible individuals who provide informed consent for participation
Attrition rate | Two weeks
  The percentage of recruited participants who did not attend the intervention or follow-up reassessment
Adherence to the intervention | Two weeks
  The percentage of sessions attended by each participant
Adverse events | Two weeks
  They will be monitored and documented after each treatment session
Accepatbility | Two weeks
  To assess the acceptability of our pilot trial and treatment process, a semi-structured interview will be conducted.

SECONDARY OUTCOMES:
Pain intensity | Two and six weeks
  11-point Numerical Pain Rating Scale, with 0 = no pain and 10 = worst pain. imaginable
Back-related disability | Two and six weeks
  The Roland Morris Disability Questionnaire consists of 24 items, with a total score of 24 and a higher score indicating greater functional limitation.
Insomnia severity | Two and six weeks
  The Insomnia Severity Index consists of seven items, with a total score of 28 and a higher score indicating severer insomnia.
Sleep quality | Two and six weeks
  The Pittsburgh Sleep Quality Index consists of 19 individual items, with a total score of 21 and a higher score indicating poorer sleep quality.
Subjetcive sleep parameters | Two weeks
  Participants will subjectively report the time of falling asleep and waking up, sleep onset latency, and quantity and duration of nighttime awakenings. Several variables will be derived from the sleep diaries, including sleep efficiency, sleep onset latency, total sleep time, and wake after sleep onset.
Objetcive sleep parameters | Two weeks
  Actigraphy will be employed to collect objective sleep parameters. The software automatically generates relevant sleep parameters involving sleep efficiency, sleep onset latency, total sleep time, wake after sleep onset.
Quantitative Sensory Testing (QST) | Two weeks
  QST will include static pain threshold (thermal, pressure, or pinprick stimulus) and dynamic pain assessments (temporal or spatial summation of pain and conditioned pain modulation).
Electroencephalography (EEG) | Two weeks
  EEG recordings will be conducted during the resting state. Power spectral density (PSD) will be computed by a Fast Fourier Transformation and quantify the amount of oscillatory activity in five frequency bands: delta (0.5-4.0Hz), theta (4.0-8.0 Hz), alpha (8.0-13.0 Hz), beta (14.0-30.0 Hz), and gamma (30.0-10.00Hz).
Pain catastrophizing | Two and six weeks
  The Pain Catastrophizing Scale (PCS) consists of 13 items with a five-point Likert scale scoring from zero (not at all) to four (always). High total scores indicate more catastrophic thoughts.

IPD SHARING:
Plan to Share IPD: No